CLINICAL TRIAL: NCT06402916
Title: The Acute Effects of Blueberries on Cognition and Mood in the Postpartum
Acronym: BLUCAMP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Daniel Lamport, Dr Daniel Lamport, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UReading BLUCAMP
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Mood; Parents; Healthy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry drink (Experimental): 46g freeze-dried wild blueberry (Vaccinium angustifolium) powder mixed with 250 ml water.
  Interventions: Dietary Supplement: Blueberry drink
- Placebo drink (Placebo Comparator): 46g placebo powder matched for macronutrients, color, and flavor mixed with 250 ml water.
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Blueberry drink — Blueberry drink equivalent to 240g fresh blueberries.
  Arms: Blueberry drink
Dietary Supplement: Placebo drink — Drink containing no active ingredient.
  Arms: Placebo drink

SUMMARY:
Blueberries are an excellent source of natural substances (flavonoids) with well-documented health benefits. Previous research has shown that consuming a serving of blueberries can improve mood in children, healthy young adults, and young adults with depressive symptoms. These results are consistent with a growing body of evidence from human and animal studies indicating that blueberries can have a beneficial effect on brain function and mental health. The postpartum period represents a challenging period whereby mood disorders such as postpartum depression become increasingly prevalent, in addition to this, mothers and fathers often report poorer cognition during this time. Therefore, it is of interest to explore whether acute blueberry supplementation can benefit mood and cognition for parents during this sensitive time.

The aim of the present study is to examine whether consuming a drink containing powdered blueberries can improve mood and cognition in parents in the 0-6 month postpartum. The design follows a randomised, double blind, placebo controlled cross over design. Participants will be invited to take part in an in-person study investigating a fruit drink on mood and cognition. Participants will come to the Nutrition-cognition lab at the Psychology department at the University of Reading for a screening session, after providing informed consent, participants will return a week later to attend a 3-hr visit during which they will receive either a blueberry or placebo drink and complete computer tasks and standardised questionnaires. Participants will then return a week later and complete the same procedure, consuming the other intervention drink.

DETAILED DESCRIPTION:
The design follows a randomised, double blind, placebo controlled cross over design. Participants will be recruited via social media, posters in the local area, and through word of mouth and email advertisements and will be invited to take part in an in-person study investigating a fruit drink on mood and cognition. Participants will come to the Nutrition-cognition lab at the Psychology department for a screening session, during the session the study will be explained by the researcher and the participant will receive the participant information sheet. If the participant is eligible and wants to take part, they will sign the consent form. Data collected at screening will include age, ethnicity, highest level of education, marital status, specific diet, income, employment, physical illnesses, psychological diagnosis, regular medications, how old their infant is, infant gender, previous children, and age of other children as well as postnatal depression, postnatal anxiety (mother's sample only), state anxiety (father's sample only) a food frequency questionnaire and anthropometric measures to determine body mass index (BMI). Participants will then complete practice versions of the cognitive tests. Office for National Statistics recommendations will be used when collecting participants demographic details of ethnicity and income.

A week later, upon arrival at the Nutrition Cognition Lab (approximately 9am) participants will be asked to note what they had for breakfast (to ensure they have the same breakfast next week for standardisation) and a researcher will ask whether they have followed the pre-session restrictions prior to coming in for the visit (see below). Participants will then complete the mood and cognitive questionnaires (listed below) and have their blood pressure taken (duration 30 min). The order of questionnaires and cognitive tasks will be kept the same throughout the study. Participants will then be randomly allocated to consume one of two interventions (blueberry drink or a similarly flavoured placebo drink). The blueberry drink consists of 46g freeze dried wild blueberry powder mixed with 250ml water, the placebo drink contains 46g placebo powder matched for sugars and vitamin C content of the blueberry powder, mixed with 250ml water. The tests will then be repeated 2 hours after consuming the drink. Participants will be able to leave the lab and have free time for the 2hrs in between testing. During the procedure, we will also request that if participants bring their infant on the day, that they also bring a partner (friend, relative or parent of infant) to care for their infant during this time so to not distract the participant during the mood and cognitive tasks. Participants will then return to the lab a week later and carry out the same procedure, though consuming the other intervention drink. After the study has been completed, participants will be debriefed and given the opportunity to ask any questions. Participants will also be reminded of their right to withdraw their data from the study if they wish. Helplines and support web links will be provided to all participants as well as encouragement for participants to contact their GP should they wish to seek support. Helplines and weblinks include Samaritans UK and PANDAS Foundation. Weblinks to NHS, MIND and the Association for Postnatal Illness.

Pre-session restrictions: Twenty-four hours before the first and second test sessions, all participants will be advised to follow a low flavonoid diet which will be advised by an information sheet provided by the researchers upon sign-up. These restrictions will be implemented as a control measure so that other dietary flavonoids do not interfere with the results of the study and researchers will check adherence to restrictions prior to the first sitting of the study. Within this 24-hour period, participants will also be asked not to drink alcohol, caffeine or take recreational drugs. Participants will also be asked to refrain from exercise and food 2 hours before and following the intervention (water will be allowed) to avoid confounding effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a biological mother or father to an infant aged 0-6 months.
* Have a good understanding of English language

Exclusion Criteria:

* Allergic to blueberries or any other Vaccinium species
* Participation in other interventional studies within the last month
* Participants with cancer, or conditions affecting the liver, heart or kidneys due to unknown effects on flavonoid metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean current affect | 2 hours post ingestion
  Assessed using scores from the Positive and Negative Affect Scale. This questionnaire has 20 items that describe some feelings and emotions. The participant needs to mark how much they are experiencing these feelings on a scale from 1-5. This produces scores of Positive Affect and Negative Affect; higher scores reflect higher positive or negative mood, respectively.

SECONDARY OUTCOMES:
Mean state anxiety | 2 hours post ingestion
  Assessed using scores from the State-Trait Anxiety Inventory- State scale. Higher scores indicate higher levels of anxiety. This questionnaire is a measure of state and trait anxiety containing 40 items in total (20 for trait; 20 for state). Only the state scale (20 items) will be used in current research to measure situational anxiety. Participants are asked to agree or disagree with anxiety-related statements on a scale of 1-4
Mean subjective mood scores | 2 hours post ingestion
  Immediate mood scale-This questionnaire contains 22 items developed to assess dynamic components of mood. Participants are asked to rate their current mood state on a continuum using 7-point Likert scales (e.g., happy-sad, distracted-focused, sleepy-alert). For each item, an integer score between 1 and 7 is derived. The total score for this scale is the sum of the scores on all 22 items.
Blood pressure | 2 hours post ingestion
  Resting systolic and diastolic blood pressure will be taken with an ambulatory blood pressure monitor. Measurements will be taken on participants left arm and the mean of three consecutive measurements will be calculated.
Mean subjective feelings | 2 hours post ingestion
  These consists of 16 dimensions of mood: Slow-Quick Witted, Tense-Relaxed, Attentive-Dreamy, Incompetent-Proficient, Happy-Sad, Antagonistic-Friendly, Interested-Bored, Withdrawn-Social. The participant is required to mark, on a line to what extent the described state is appropriate to them at that moment in time. The individual responses from the 16 mood scales are combined to make three affective dimensions of alertness, contentment, and calmness.
Verbal memory | 2 hours post ingestion
  Assessed using the Rey Auditory Verbal Learning Test.
Sustained attention and executive functioning | 2 hours post ingestion
  Assessed with the Modified Attention Network Task with accuracy and reaction time as outcome measures.
Visuospatial working memory | 2 hours post ingestion
  Measured using the Visuospatial n-back with accuracy and reaction time as outcome measures.

OTHER OUTCOMES:
General diet | Screening
  Participants will complete a food frequency questionnaire at baseline using the EPIC FFQ. This measures contains a list of foods/drinks and the participant needs to state how often they consume each food/drink to assess participants' general diet.
Subjective sleep scores | Baseline
  Using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a validated measure of sleep assessing qualities and patterns within the last month of sleep habits in adults. Seven components of sleep (quality, latency, duration, efficiency, disturbance, use of sleep medication, daytime dysfunction) will be summed to achieve a global PSQI score ranging from 0 to 21 points, where scores above 5 indicates sleep problems.
Mean postpartum-specific anxiety symptoms | Screening
  Assessed using scores from the Postpartum-Specific Anxiety Scale. This is a 51-item questionnaire that examines the frequency of maternal and infant focused anxieties experienced by women over the last week. It can be used at any time during the first year following birth and is found to be a valid and reliable measure. Each response is given a score of between 1 and 4 with the maximum score being a total of 204, with higher scores indicating higher levels of anxiety where a score of 112 or above indicating likelihood the individual suffering from an anxiety disorder. As this is maternal specific, the questionnaire will only be given to the mothers sample.
Mean trait anxiety | Screening
  Assessed using scores from the State-Trait Anxiety Inventory- trait scale. Higher scores indicate higher levels of anxiety. This questionnaire is a measure of state and trait anxiety containing 40 items in total (20 for trait; 20 for state). Only the trait scale (20 items) will be used in current research to measure trait anxiety. Participants are asked to agree or disagree with anxiety-related statements on a scale of 1-4. This questionnaire will only be used in the fathers sample to measure fathers anxiety.
Mean depressive symptoms | Screening
  Assessed using scores from the Edinburgh Postnatal Depression Scale measure. Higher scores indicate higher levels of depressive symptoms. This questionnaire contains 10 items where participants rate how they have been feeling over the past 7 days on a 4-point Likert scale. The EPDS was designed for women who are pregnant or have just had a baby and has shown to be an efficient and effective way of identifying patients at risk for perinatal depression. This measure is suitable for use in new mothers and fathers.
Mean subjective stress scores | Baseline
  Measures using the Percieved Stress Scale designed to measure stress in the last month. Participants are asked to rate their feelings on a continuum using 5-point Likert scales from 0 (never) to 4 (very often). The total score for this questionnaire is 40 with higher scores indicating more stress.
Drink rating scale | Immediately post ingestion
  Participants will be asked to rate 8 questions on a scale of 0-9 how palatable the intervention drinks are.
Mean overall infant temperament scores | Screening
  This questionnaire explores early infant temperament and asks parents to rate their infants temperament in the last 7 days. For the purpose of this study, only the 'Overall impressions and experiences subscale' will be used which explores 'Easiness of baby' and 'Global confidence'. This particular subscale consists of seven questions which are rated on seven-point scales from '-3' to '+3', with -3 signifying 'very difficult' behaviours and +3 'very easy' ones (e.g. -3 = 'very irritable'/ +3 = 'very calm'). The total score will be taken, with lower scores representing a more irritable infant.
Mean daily infant temperament scores | Baseline
  This questionnaire explores early infant temperament and asks parents to rate their infants temperament in the last 7 days. For the purpose of this study, only the 'Overall impressions and experiences subscale' will be used which explores 'Easiness of baby' and 'Global confidence'. This particular subscale consists of seven questions which are rated on seven-point scales from '-3' to '+3', with -3 signifying 'very difficult' behaviours and +3 'very easy' ones (e.g. -3 = 'very irritable'/ +3 = 'very calm'). The first question on the scale "How irritable is your baby" will be used at each test day to understand their infants temperament at the visit.
Mean subjective memory scores | Screening
  Prospective and retrospective memory questionnaire. The PRMQ is a 16-item rating scale, designed to assess the frequency of different types of memory failures whereby higher scores indicate greater frequency of memory failures. Participants are asked to score questions of a 5-point scale 1 (never), 2 (rarely), 3 (sometimes), 4 (quite often), 5 (very often). Results can be derived for prospective or retrospective, short-term or long-term, self-cued or environmentally cued.

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data may be made available on a platform such as Open Science Framework (www.osf.io) or a data repository linked to academic journals, in accordance with Open Science principles.